CLINICAL TRIAL: NCT01444534
Title: Influence of a Mobile Phone Application on Quality of Life of Patients With Type 1 Diabetes Mellitus: a Randomized Controlled Trial
Brief Title: Mobile Phone Applications and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Research Foundation, The Netherlands (Other)
Responsible Party: Principal Investigator, Nanne Kleefstra, ass. professor, Medical Research Foundation, The Netherlands
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pameijer-2011
Record Dates: First submitted 2011-09-26; First posted 2011-09-30 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Type 1 Diabetes
Keywords: mobile phone application; diabetes type 1; self-management; telemedicin
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- use of the diabetes application (Experimental)
  Interventions: Device: Dbees; diabetes mobile phone application
- Control arm without app (usual care) (Active Comparator)
  Interventions: Device: control group

INTERVENTIONS:
Device: Dbees; diabetes mobile phone application — Participants randomized to the intervention group (G2) were asked to stop using their paper logbook and start using an electronic logbook on their computer and mobile phone using an application of Dbees. The Dbees software enables the mobile phone to be used as a small computer to record the blood glucose values, dose of insulin injection, daily carbohydrate intake, amount of physical activity, and blood pressure.
  Arms: use of the diabetes application
Device: control group — Participants in the control group (G1) continued using their paper logbook (usual care) and had no electronic logbook. Patients in the control group were requested not to use another mobile phone application instead of or besides their paper logbook.
  Arms: Control arm without app (usual care)

SUMMARY:
The use of smartphones has increased substantially in recent years. Apart from making phone calls and sending short messages, these smartphones can also function as a computer on which one can download computer programs (the so-called applications). Health applications are increasingly developed and may be a new tool for education of patients and communication between healthcare providers and their patients, possibly contributing to a better care for patients with chronic diseases such as diabetes.

Since the number of patients with diabetes mellitus and the number of people having a smartphone are rising, it is investigated whether applications on smartphones may be used to support lifestyle changes and self-monitoring of bloodglucose control, possibly leading to an improved glycaemic regulation in the group of patients with diabetes mellitus.

Large randomized controlled trials have shown that a stable glycaemic regulation is important to reduce morbidity and mortality and to improve quality of life (QOL). Self-monitoring of blood glucose is an important tool to realize an optimal glycaemic regulation in patients with type 1 diabetes mellitus (T1DM). Apart from a good glycaemic control, QOL is essential in diabetic patients. A reduced QOL is associated with progression of the disease, worse intake of medication and an increased mortality in patients with T1DM and diabetes mellitus type 2.

The increasing costs associated with the rising number of diabetic patients makes that research investigating cheaper alternatives in the care for patients with diabetes are needed. The switch from a written logbook to an electronic logbook may simplify the care for diabetes patients. By means of an application all variables (food intake, physical exercise, glucose day curves, insulin units, reminders to take medication) are integrated in one program. But whether this digitalisation also improves QOL of the patient is still unclear.

Therefore the aim of this study is to evaluate the effect of a diabetes application on the (QOL) for type 1 diabetic patients.

DETAILED DESCRIPTION:
Participants in both groups were invited to participate after their periodical visit to the doctor or the hospital-based nurse specialised in the care for diabetes patients. All participants in this study were adults with T1DM having a smartphone.

All participants will complete the The Short Form Health Survey (SF-36) and the Problem Areas In Diabetes questionnaire (PAID) at baseline and after three months of follow-up. Baseline information, including socio demographic information (age, sex, highest level of school education), and clinical characteristics (diabetes duration, insulin therapy and presence and severity of diabetes complications) will be collected in a database. Moreover parameters such as blood pressure, body weight, HbA1c and lipid profile will be added.

Sample size calculation

The study was powered to detect a between-group mean difference of 10 points in the The Short Form Health Survey (SF-36) questionnaire after 3 months. With a power of 80%, alpha 0.05, the total sample size of the study should be 62 patients (31 in each group).

ELIGIBILITY:
Inclusion Criteria:

* diabetes type 1
* >18 years old
* patient having a smartphone, who are familiar with its use

Exclusion Criteria:

* previous or actual use of a diabetes application
* pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2011-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 3 months

SECONDARY OUTCOMES:
HbA1c | 3 months
usability of the application | 3 months
  questionnaire System Usability Scale (SUS)
Self-monitoring of blood glucose (SMBG) | 3 months
  frequency of blood glucose monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Henk J. Bilo, MD/PhD, Principal Investigator — Isala clinics, medical research foundation
Locations (1):
- Isala Clinics, Zwolle, Netherlands